CLINICAL TRIAL: NCT02462187
Title: A Phase 2, Multi-center, Double-blind, Randomized, Vehicle-controlled, Ascending Dose Study Assessing Tolerability, Safety, and Efficacy of Topical NVN1000 in Subjects With External Genital Warts and Perianal Warts
Brief Title: Topical NVN1000 for the Treatment of External Genital and Perianal Warts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novan, Inc. (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NI-WA201
Record Dates: First submitted 2015-05-28; First posted 2015-06-03 (Estimated); Results first posted 2023-04-05 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Genital Warts; Perianal Warts
Keywords: genital warts; perianal warts
MeSH Terms: conditions — Condylomata Acuminata | interventions — berdazimer sodium; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- NVN1000 8% Gel twice daily (Experimental): NVN1000 8% Gel twice daily
  Interventions: Drug: NVN1000 8% Gel
- NVN1000 8% Gel once daily (Experimental): NVN1000 8% Gel once daily
  Interventions: Drug: NVN1000 8% Gel
- NVN1000 16% Once daily (Experimental): NVN1000 16% Gel once daily
  Interventions: Drug: NVN1000 16%
- Vehicle Gel (Placebo Comparator): Vehicle Gel at frequency to match active
  Interventions: Drug: Vehicle
- NVN1000 24% once daily (Experimental): NVN1000 24% once daily
  Interventions: Drug: NVN1000 24%

INTERVENTIONS:
Drug: NVN1000 8% Gel — once and twice daily
  Other Names: SB206
  Arms: NVN1000 8% Gel once daily; NVN1000 8% Gel twice daily
Drug: NVN1000 16% — once daily
  Other Names: SB206
  Arms: NVN1000 16% Once daily
Drug: Vehicle — placebo comparator
  Other Names: Placebo
  Arms: Vehicle Gel
Drug: NVN1000 24% — once daily
  Other Names: SB206
  Arms: NVN1000 24% once daily

SUMMARY:
A Phase 2 Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Ascending Dose Study Assessing Tolerability, Safety, and Efficacy of Topical NVN1000 in Subjects with External Genital Warts and Perianal Warts

DETAILED DESCRIPTION:
This is a phase 2, multi-center, randomized, double-blind, vehicle-controlled, ascending dose study to assess safety, tolerability and efficacy of a topical nitric oxide releasing compound in subjects with external genital and perianal warts. Eligible subjects will be treated with a topical gel (active or vehicle) for up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 but not more than 20 genital/perianal warts with a maximum total wart surface area no more than 1% body surface area
* If a woman of child-bearing potential, have a negative pregnancy test and use effective contraception
* If currently receiving wart treatment, be willing to stop all treatment for 28 days prior to randomization and during the study

Exclusion Criteria:

* Immunocompromised patients including those with HIV, receiving radiation, or drugs that suppress the immune system
* Pregnant, planning to become pregnant, or nursing
* History of cancer (including cervical cancer) within 5 years, with exception of non-melanoma skin cancer in non-genital skin
* Recent history of other genital skin infections
* Active HSV and frequent HSV recurrences unless receiving suppression therapy
* Have hemoglobin < 10 G/dl or methemoglobin > 3%
* Known allergy to any component of the gel including excipients
* Previously participated in any study with NVN1000 or SB204

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2015-06-12 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Rico, MD, Study Director — Novan, Inc.
Locations (15):
- United States (15):
  - PPD 137, Fountain Valley, California
  - PPD 140, Lomita, California
  - PPD 133, San Diego, California
  - PPD 134, Atlanta, Georgia
  - PPD 139, Atlanta, Georgia
  - PPD 138, Roswell, Georgia
  - PPD 130, Indianapolis, Indiana
  - PPD 126, Metairie, Louisiana
  - PPD 132, Portland, Oregon
  - PPD 135, Philadelphia, Pennsylvania
  - PPD 128, Corpus Christi, Texas
  - PPD 129, Houston, Texas
  - PPD 127, San Antonio, Texas
  - PPD 131, Webster, Texas
  - PPD 136, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 120 subjects were planned to be enrolled; 108 subjects were actually enrolled per the Sponsor's decision.
Groups:
- Cohort 1: NVN1000 8% Gel Twice Daily: NVN1000 8% Gel applied topically twice daily
- Cohort 2: NVN1000 8% Gel Once Daily: NVN1000 8% Gel applied topically once daily
- Cohort 3: NVN1000 16% Once Daily: NVN1000 16% Gel applied topically once daily
- Cohort 4: NVN1000 24% Once Daily: NVN1000 24% applied topically once daily
- Vehicle Gel Once Daily; Vehicle Gel Twice Daily: Vehicle: placebo comparator
Period: Overall Study
Arm/Group | Cohort 1: NVN1000 8% Gel Twice Daily | Cohort 2: NVN1000 8% Gel Once Daily | Cohort 3: NVN1000 16% Once Daily | Cohort 4: NVN1000 24% Once Daily | Vehicle Gel Once Daily | Vehicle Gel Twice Daily
Started | 13 | 24 | 14 | 30 | 23 | 4
Completed | 8 | 19 | 9 | 23 | 16 | 4
Not Completed | 5 | 5 | 5 | 7 | 7 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat Population (ITT)--the ITT includes all study subjects who were randomized and dispensed study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: NVN1000 8% Gel Twice Daily | Cohort 2: NVN1000 8% Gel Once Daily | Cohort 3: NVN1000 16% Once Daily | Cohort 4: NVN1000 24% Once Daily | Vehicle Gel Once Daily | Vehicle Gel Twice Daily | Total
Number analyzed (Participants) | 12 | 24 | 14 | 30 | 23 | 4 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (7.13) | 33.3 (6.68) | 32.5 (7.86) | 33.6 (6.77) | 32.2 (7.41) | 31.5 (9.00) | 33.4 (7.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 2 | 7 | 6 | 2 | 31
  Male | 6 | 16 | 12 | 23 | 17 | 2 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 5 | 5 | 9 | 2 | 30
  Not Hispanic or Latino | 9 | 18 | 9 | 25 | 14 | 2 | 77
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 8 | 3 | 10 | 5 | 0 | 29
  White | 9 | 16 | 11 | 19 | 17 | 4 | 76
  More than one race | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 24 | 14 | 30 | 23 | 4 | 107
Current Tobacco Use [Count of Participants; unit: Participants]
  Yes | 5 | 5 | 2 | 12 | 8 | 3 | 35
  No | 7 | 19 | 12 | 18 | 15 | 1 | 72
Wart Location at Baseline [Count of Participants; unit: Participants]
  External genital warts (EGW) only | 9 | 17 | 13 | 19 | 15 | 3 | 76
  Perianal warts (PAW) only | 2 | 2 | 0 | 7 | 1 | 1 | 13
  EGW and PAW | 1 | 5 | 1 | 4 | 7 | 0 | 18
Baseline Wart Count [Mean (Standard Deviation); unit: number of warts] | 9.3 (5.93) | 7.5 (5.05) | 5.1 (2.60) | 7.2 (5.58) | 7.7 (5.83) | 7.8 (3.40) | 7.4 (5.19)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Complete Clearance of Baseline External Genital and Perianal Warts at or Before Week 12
Description: Clearance of baseline external genital and perianal warts at or before Week 12 as determined by physical examination by the investigator.
Time Frame: 12 weeks
Population: ITT population. One subject in the NVN1000 8% Gel BID group was randomized but not dispensed treatment and thus was excluded from the ITT population..
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: NVN1000 8% Gel Twice Daily | Cohort 2: NVN1000 8% Gel Once Daily | Cohort 3: NVN1000 16% Once Daily | Cohort 4: NVN1000 24% Once Daily | Vehicle Gel Once Daily | Vehicle Gel Twice Daily
Number analyzed (Participants) | 12 | 24 | 14 | 30 | 23 | 4
Participants | 2 | 5 | 2 | 10 | 1 | 2

2. Secondary Outcome: Tolerability of Topical NVN1000 Gel as Determined by Scores on a 4 Point Grading Scale for Erythema, Edema, Erosions/Ulcers, and Itch
Description: Comparison of scores for erythema, edema, erosions/ulcers, itch between active and vehicle treated subjects using a 4 point grading scale; on the tolerability scale, 0 = none and 3 = severe, indicating an increase in severity the higher the number assigned.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: NVN1000 8% Gel Twice Daily | Cohort 2: NVN1000 8% Gel Once Daily | Cohort 3: NVN1000 16% Once Daily | Cohort 4: NVN1000 24% Once Daily | Vehicle Gel Once Daily | Vehicle Gel Twice Daily
Number analyzed (Participants) | 12 | 23 | 14 | 30 | 20 | 4
Participants
  Erythema: Baseline: 0 (none) | 12 | 23 | 14 | 27 | 20 | 4
  Erythema: Baseline: 1 (mild) | 0 | 0 | 0 | 2 | 0 | 0
  Erythema: Baseline: 2 (moderate) | 0 | 0 | 0 | 0 | 0 | 0
  Erythema: Baseline: 3 (severe) | 0 | 0 | 0 | 0 | 0 | 0
  Erythema: Baseline: Missing/unknown | 0 | 0 | 0 | 1 | 0 | 0
  Erythema: Week 2: 0 (none) | 6 | 16 | 11 | 19 | 18 | 4
  Erythema: Week 2: 1 (mild) | 2 | 4 | 1 | 9 | 1 | 0
  Erythema: Week 2: 2 (moderate) | 3 | 2 | 2 | 2 | 0 | 0
  Erythema: Week 2: 3 (severe) | 1 | 0 | 0 | 0 | 0 | 0
  Erythema: Week 2: Missing/unknown | 0 | 1 | 0 | 0 | 1 | 0
  Erythema: Week 4: 0 (none) | 6 | 14 | 9 | 20 | 19 | 4
  Erythema: Week 4: 1 (mild) | 3 | 4 | 3 | 6 | 0 | 0
  Erythema: Week 4: 2 (moderate) | 0 | 3 | 1 | 2 | 0 | 0
  Erythema: Week 4: 3 (severe) | 0 | 0 | 0 | 0 | 0 | 0
  Erythema: Week 4: Missing/unknown | 3 | 2 | 1 | 2 | 1 | 0
  Erythema: Week 8: 0 (none) | 8 | 13 | 8 | 18 | 16 | 4
  Erythema: Week 8: 1 (mild) | 0 | 3 | 2 | 3 | 1 | 0
  Erythema: Week 8: 2 (moderate) | 1 | 2 | 1 | 4 | 0 | 0
  Erythema: Week 8: 3 (severe) | 0 | 0 | 0 | 1 | 0 | 0
  Erythema: Week 8: Missing/unknown | 3 | 5 | 3 | 4 | 3 | 0
  Erythema: Week 12: 0 (none) | 8 | 15 | 6 | 19 | 18 | 4
  Erythema: Week 12: 1 (mild) | 0 | 2 | 2 | 3 | 2 | 0
  Erythema: Week 12: 2 (moderate) | 0 | 2 | 1 | 0 | 0 | 0
  Erythema: Week 12: 3 (severe) | 0 | 0 | 0 | 1 | 0 | 0
  Erythema: Week 12: Missing/unknown | 4 | 4 | 5 | 7 | 0 | 0
  Edema: Baseline: 0 (none) | 12 | 23 | 14 | 28 | 20 | 4
  Edema: Baseline: 1 (mild) | 0 | 0 | 0 | 1 | 0 | 0
  Edema: Baseline: 2 (moderate) | 0 | 0 | 0 | 0 | 0 | 0
  Edema: Baseline: 3 (severe) | 0 | 0 | 0 | 0 | 0 | 0
  Edema: Baseline: Missing/unknown | 0 | 0 | 0 | 1 | 0 | 0
  Edema: Week 2: 0 (none) | 10 | 22 | 12 | 26 | 19 | 4
  Edema: Week 2: 1 (mild) | 0 | 0 | 1 | 4 | 0 | 0
  Edema: Week 2: 2 (moderate) | 2 | 0 | 1 | 0 | 0 | 0
  Edema: Week 2: 3 (severe) | 0 | 0 | 0 | 0 | 0 | 0
  Edema: Week 2: Missing/unknown | 0 | 1 | 0 | 0 | 1 | 0
  Edema: Week 4: 0 (none) | 9 | 19 | 11 | 25 | 19 | 4
  Edema: Week 4: 1 (mild) | 1 | 2 | 2 | 3 | 0 | 0
  Edema: Week 4: 2 (moderate) | 0 | 0 | 0 | 0 | 0 | 0
  Edema: Week 4: 3 (severe) | 0 | 0 | 0 | 0 | 0 | 0
  Edema: Week 4: Missing/unknown | 2 | 2 | 1 | 2 | 1 | 0
  Edema: Week 8: 0 (none) | 8 | 18 | 10 | 24 | 17 | 4
  Edema: Week 8: 1 (mild) | 1 | 0 | 0 | 1 | 0 | 0
  Edema: Week 8: 2 (moderate) | 0 | 0 | 1 | 1 | 0 | 0
  Edema: Week 8: 3 (severe) | 0 | 0 | 0 | 0 | 0 | 0
  Edema: Week 8: Missing/unknown | 3 | 5 | 3 | 4 | 3 | 0
  Edema: Week 12: 0 (none) | 8 | 18 | 8 | 20 | 16 | 4
  Edema: Week 12: 1 (mild) | 0 | 1 | 1 | 2 | 0 | 0
  Edema: Week 12: 2 (moderate) | 0 | 0 | 0 | 1 | 0 | 0
  Edema: Week 12: 3 (severe) | 0 | 0 | 0 | 0 | 0 | 0
  Edema: Week 12: Missing/unknown | 4 | 4 | 5 | 7 | 4 | 0
  Erosion/Ulceration: Baseline: 0 (none) | 12 | 23 | 14 | 28 | 20 | 4
  Erosion/Ulceration: Baseline: 1 (mild) | 0 | 0 | 0 | 1 | 0 | 0
  Erosion/Ulceration: Baseline: 2 (moderate) | 0 | 0 | 0 | 0 | 0 | 0
  Erosion/Ulceration: Baseline: 3 (severe) | 0 | 0 | 0 | 0 | 0 | 0
  Erosion/Ulceration: Baseline: Missing/unknown | 0 | 0 | 0 | 1 | 0 | 0
  Erosion/Ulceration: Week 2: 0 (none) | 8 | 18 | 14 | 27 | 19 | 4
  Erosion/Ulceration: Week 2: 1 (mild) | 3 | 4 | 0 | 2 | 0 | 0
  Erosion/Ulceration: Week 2: 2 (moderate) | 0 | 0 | 0 | 0 | 0 | 0
  Erosion/Ulceration: Week 2: 3 (severe) | 1 | 0 | 0 | 1 | 0 | 0
  Erosion/Ulceration: Week 2: Missing/unknown | 0 | 1 | 0 | 0 | 1 | 0
  Erosion/Ulceration: Week 4: 0 (none) | 9 | 18 | 13 | 24 | 19 | 4
  Erosion/Ulceration: Week 4: 1 (mild) | 0 | 2 | 0 | 3 | 0 | 0
  Erosion/Ulceration: Week 4: 2 (moderate) | 1 | 0 | 0 | 1 | 0 | 0
  Erosion/Ulceration: Week 4: 3 (severe) | 0 | 1 | 0 | 0 | 0 | 0
  Erosion/Ulceration: Week 4: Missing/unknown | 2 | 2 | 1 | 2 | 1 | 0
  Erosion/ulceration: Week 8: 0 (none) | 8 | 15 | 11 | 20 | 20 | 4
  Erosion/ulceration: Week 8: 1 (mild) | 0 | 2 | 0 | 4 | 0 | 0
  Erosion/ulceration: Week 8: 2 (moderate) | 1 | 1 | 0 | 2 | 0 | 0
  Erosion/ulceration: Week 8: 3 (severe) | 0 | 0 | 0 | 0 | 0 | 0
  Erosion/ulceration: Week 8: Missing/unknown | 3 | 5 | 3 | 4 | 0 | 0
  Erosion/ulceration: Week 12: 0 (none) | 8 | 16 | 8 | 20 | 20 | 4
  Erosion/ulceration: Week 12: 1 (mild) | 0 | 3 | 1 | 2 | 0 | 0
  Erosion/ulceration: Week 12: 2 (moderate) | 0 | 0 | 0 | 1 | 0 | 0
  Erosion/ulceration: Week 12: 3 (severe) | 0 | 0 | 0 | 0 | 0 | 0
  Erosion/ulceration: Week 12: Missing/unknown | 4 | 4 | 5 | 7 | 0 | 0
  Burning/stinging: Baseline: 0 (none) | 12 | 23 | 14 | 28 | 20 | 4
  Burning/stinging: Baseline: 1 (mild) | 0 | 0 | 0 | 0 | 0 | 0
  Burning/stinging: Baseline: 2 (moderate) | 0 | 0 | 0 | 1 | 0 | 0
  Burning/stinging: Baseline: 3 (severe) | 0 | 0 | 0 | 0 | 0 | 0
  Burning/stinging: Baseline: Missing/unknown | 0 | 0 | 0 | 1 | 0 | 0
  Burning/stinging: Week 2: 0 (none) | 6 | 16 | 8 | 17 | 15 | 2
  Burning/stinging: Week 2: 1 (mild) | 3 | 5 | 4 | 10 | 4 | 2
  Burning/stinging: Week 2: 2 (moderate) | 0 | 1 | 2 | 3 | 0 | 0
  Burning/stinging: Week 2: 3 (severe) | 3 | 0 | 0 | 0 | 0 | 0
  Burning/stinging: Week 2: Missing/unknown | 0 | 1 | 0 | 0 | 1 | 0
  Burning/stinging: Week 4: 0 (none) | 6 | 15 | 6 | 18 | 16 | 3
  Burning/stinging: Week 4: 1 (mild) | 2 | 3 | 7 | 5 | 3 | 1
  Burning/stinging: Week 4: 2 (moderate) | 2 | 3 | 0 | 2 | 0 | 0
  Burning/stinging: Week 4: 3 (severe) | 0 | 0 | 0 | 3 | 0 | 0
  Burning/stinging: Week 4: Missing/unknown | 2 | 2 | 1 | 2 | 1 | 0
  Burning/stinging: Week 8: 0 (none) | 6 | 13 | 8 | 19 | 13 | 2
  Burning/stinging: Week 8: 1 (mild) | 1 | 3 | 2 | 6 | 3 | 2
  Burning/stinging: Week 8: 2 (moderate) | 2 | 2 | 1 | 1 | 1 | 0
  Burning/stinging: Week 8: 3 (severe) | 0 | 0 | 0 | 0 | 0 | 0
  Burning/stinging: Week 8: Missing/unknown | 3 | 5 | 3 | 4 | 3 | 0
  Burning/stinging: Week 12: 0 (none) | 6 | 13 | 8 | 19 | 14 | 4
  Burning/stinging: Week 12: 1 (mild) | 1 | 3 | 1 | 2 | 1 | 0
  Burning/stinging: Week 12: 2 (moderate) | 1 | 3 | 0 | 1 | 1 | 0
  Burning/stinging: Week 12: 3 (severe) | 0 | 0 | 0 | 1 | 0 | 0
  Burning/stinging: Week 12: Missing/unknown | 4 | 4 | 5 | 7 | 4 | 0

3. Secondary Outcome: Safety as Determined by Changes in Laboratory Assessments
Description: Safety population--Comparison of changes in methemoglobin levels between active and vehicle treated subjects. Methemoglobin levels were measured using a RAD-57 pulse co-oximeter. Values are expressed as a percentage of hemoglobin.
Time Frame: Baseline, Week 2 and Week 12
Population: Safety population
Measure: Mean (Full Range); unit: Percentage
Arm/Group | Cohort 1: NVN1000 8% Gel Twice Daily | Cohort 2: NVN1000 8% Gel Once Daily | Cohort 3: NVN1000 16% Once Daily | Cohort 4: NVN1000 24% Once Daily | Vehicle Gel Once Daily | Vehicle Gel Twice Daily
Number analyzed (Participants) | 12 | 23 | 14 | 30 | 20 | 4
Percentage
  Baseline | 1.33 [0.7 to 1.7] | 1.25 [0.7 to 2.1] | 1.38 [0.8 to 2.1] | 1.29 [0.6 to 2.1] | 1.31 [0.5 to 2.0] | 1.53 [1.2 to 1.7]
  Week 2: number analyzed (Participants) | 12 | 22 | 14 | 30 | 19 | 4
  Week 2 | 1.33 [0.7 to 2.0] | 1.33 [0.9 to 2.7] | 1.42 [0.9 to 1.9] | 1.33 [0.8 to 2.1] | 1.34 [0.9 to 1.9] | 1.48 [1.2 to 1.7]
  Week 12: number analyzed (Participants) | 10 | 19 | 10 | 25 | 16 | 4
  Week 12 | 1.55 [1.0 to 2.5] | 1.34 [0.8 to 2.8] | 1.26 [0.8 to 1.8] | 1.36 [0.9 to 2.1] | 1.59 [0.7 to 4.0] | 1.50 [1.1 to 2.7]

4. Secondary Outcome: Percentage of Subjects With Complete Clearance of Total EGW/PAW at or Before Week 12
Description: The percentage of subjects with complete clearance of baseline and warts that emerge during treatment period as determined by physical examination by the investigator
Time Frame: 12 weeks
Population: Intent to treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: NVN1000 8% Gel Twice Daily | Cohort 2: NVN1000 8% Gel Once Daily | Cohort 3: NVN1000 16% Once Daily | Cohort 4: NVN1000 24% Once Daily | Vehicle Gel Once Daily | Vehicle Gel Twice Daily
Number analyzed (Participants) | 12 | 24 | 14 | 30 | 23 | 4
Participants | 2 | 5 | 2 | 9 | 1 | 2

5. Secondary Outcome: Percentage of Subjects With Complete or Partial Clearance of Baseline Warts at or Before Week 12
Description: Percentage of subjects with complete or partial clearance of baseline warts as determined by physical examination by the investigator
Time Frame: 12 weeks
Population: Intent to treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: NVN1000 8% Gel Twice Daily | Cohort 2: NVN1000 8% Gel Once Daily | Cohort 3: NVN1000 16% Once Daily | Cohort 4: NVN1000 24% Once Daily | Vehicle Gel Once Daily | Vehicle Gel Twice Daily
Number analyzed (Participants) | 12 | 24 | 14 | 30 | 23 | 4
Participants | 8 | 19 | 10 | 17 | 11 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject signed the informed consent and completed any study assessment until the end of the final study visit, up to approximately 12 weeks.
Description: Safety population: The safety population included all randomized subjects with documented use of study medication (at least one application) at at least one post-baseline safety assessment.
Arm/Group | Cohort 1: NVN1000 8% Gel Twice Daily | Cohort 2: NVN1000 8% Gel Once Daily | Cohort 3: NVN1000 16% Once Daily | Cohort 4: NVN1000 24% Once Daily | Vehicle Gel Once Daily | Vehicle Gel Twice Daily
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/23 | 0/14 | 0/30 | 0/20 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/12 | 0/23 | 1/14 | 0/30 | 0/20 | 0/4
Other Adverse Events (participants affected / at risk) | 9/12 | 13/23 | 5/14 | 7/30 | 4/20 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: NVN1000 8% Gel Twice Daily (N=12) | Cohort 2: NVN1000 8% Gel Once Daily (N=23) | Cohort 3: NVN1000 16% Once Daily (N=14) | Cohort 4: NVN1000 24% Once Daily (N=30) | Vehicle Gel Once Daily (N=20) | Vehicle Gel Twice Daily (N=4)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: NVN1000 8% Gel Twice Daily (N=12) | Cohort 2: NVN1000 8% Gel Once Daily (N=23) | Cohort 3: NVN1000 16% Once Daily (N=14) | Cohort 4: NVN1000 24% Once Daily (N=30) | Vehicle Gel Once Daily (N=20) | Vehicle Gel Twice Daily (N=4)
Application Site Burn (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application Site Erosion (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Application Site Erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Application Site Exfoliation (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application Site Pain (General disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (6) | 0 (0) | 0 (0)
Application Site Pruritus (General disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application Site Rash (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application Site Reaction (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Application Site Ulcer (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Viral Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Affective Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-03-22): https://cdn.clinicaltrials.gov/large-docs/87/NCT02462187/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/87/NCT02462187/SAP_001.pdf